CLINICAL TRIAL: NCT04360460
Title: Role of Functional Translation After Immersive Virtual Reality Exposure in Persons With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5200147
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Hemiparesis as Late Effect of Cerebrovascular Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Virtual reality followed by translation into related functional tasks in a real life setting for 2 weeks + conventional therapies
  Interventions: Other: Immersive virtual reality + related functional translation into real-life
- Control (Active Comparator): Virtual reality followed by translation into non-related functional tasks in a real life setting for 2 weeks + conventional therapies
  Interventions: Other: Immersive virtual reality + non-related translation into real-life

INTERVENTIONS:
Other: Immersive virtual reality + related functional translation into real-life — The experimental group will perform tasks in an immersive virtual reality setting designed to encourage functional task performance for 30 minutes. The patient will then be brought to a real-life setting and evaluated on similar task performances for an additional 30 minutes for a total of 60 minutes per day, 3 times a week for 2 weeks.
  Arms: Experimental
Other: Immersive virtual reality + non-related translation into real-life — The control group will also be asked to perform tasks in an immersive VR setting for 30 minutes, however tasks will be unrelated to the tasks performed in the real-life setting in the following 30 minutes. The control group will also receive 60 minutes of therapy a day, 3 times a week, for 2 weeks.
  Arms: Control

SUMMARY:
This is a single-blinded randomized control trial aiming to explore the use of immersive virtual reality (VR) training in conjunction with real-life tasks therapy in 75 first time stroke patients with upper limb weakness.

DETAILED DESCRIPTION:
Patients will be randomized to a control or experimental group. The experimental group will receive immersive VR training followed by the translation of related tasks in a real life environment. The control group will perform the same tasks in a real life environment but will receive immersive VR exposure to a non-related task.

ELIGIBILITY:
Inclusion Criteria:

1. 18-90 years old
2. Hospitalized at Loma Linda East Campus Rehabilitation Hospital
3. First time stroke patient
4. Upper limb hemiparesis
5. English-speaking
6. Manual muscle testing of at least 2/5 in 3 or more muscle groups in affected upper limb

Exclusion Criteria:

1. Active neck pain, headaches, or vertigo limiting ability to tolerate Virtual Reality Head Mounted Device
2. Patients with hemicraniectomy
3. Current uncontrolled seizures
4. Active infections requiring contact precautions
5. Cognitively unable to participate
6. Vision loss limiting ability to participate with VR therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Motor Activity Log | Change in score (between baseline and time of discharge from rehabilitation hospital, about 2 weeks)
  ADL Self-Reported Questionnaire
  Amount Scale (0-5) 0 = Did not use my weaker arm (not used) 5 = Used my weaker arm as often as before the stroke (same as pre-stroke).
  How well scale (0-5) 0 - My weaker arm was not used at all for that activity (not used). 5 - The ability to use my weaker arm for that activity was as good as before the stroke (normal).

SECONDARY OUTCOMES:
Modified Barthel's Index | Change in score (between baseline and time of discharge from rehabilitation hospital, about 2 weeks)
  Quality of Life Self-Reported Questionnaire
  80-100 Independent 60-79 Minimally dependent 40-59 Partially dependent 20-39 Very dependent <20 Totally dependent
Fugl-Meyer Upper Extremity Assessment | Change in score (between baseline and time of discharge from rehabilitation hospital, about 2 weeks)
  Post-stroke upper extremity assessment
  Very severe = 0-35 Severe = 36-55 Moderate. = 56-79 Slight = >79
Montreal Cognitive Assessment | Change in score (between baseline and time of discharge from rehabilitation hospital, about 2 weeks)
  Cognitive Assessment
  No cognitive impairment: MoCA ≥ 25 Mild cognitive impairment: MoCA 20-24 Severe cognitive impairment: MoCA < 20
Functional Independence Measurement Score | Change in score (between baseline and time of discharge from rehabilitation hospital, about 2 weeks)
  Functional evaluation
  7 - complete independence 6 - modified indepdendence 5 - supervision/Setup 4 - minimal contact assistance 3 - moderate assistance 2 - maximal assistance
  1 - total assistance 0 - activity does not occur

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tarver, MD, Principal Investigator — Loma Linda University
Locations (1):
- Tom and Vi Zapara Rehabilitation Pavilion, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No